CLINICAL TRIAL: NCT00079534
Title: Distant Healing Efforts for AIDS by Nurses and "Healers"
Brief Title: Distant Healing for HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000485-01 (NIH)
Record Dates: First submitted 2004-03-09; First posted 2004-03-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections; AIDS
Keywords: AIDS; HIV; Prayer; Healing; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: Non-local/distant healing or prayer

SUMMARY:
The purpose of this study is to determine whether individuals praying at a distance (also known as "Distant Healing") can positively affect the health of people with HIV/AIDS.

DETAILED DESCRIPTION:
Significant numbers of people with HIV/AIDS seek spiritual or "psychic" treatment. Distant healing could potentially be of benefit to large numbers of HIV/AIDS patients, as it is widely available and requires no travel or other activity on the part of the patient. However, the treatment can be costly and has not yet been proven effective in a controlled clinical trial. This study will evaluate the efficacy of distant healing in patients with HIV/AIDS.

Participants in this study will be randomly assigned to either the distant healing group or a control group. All participants will have hour-long study visits at entry and Months 6 and 12. At study visits, participants will complete a demographic questionnaire, self-report health and symptom inventory, quality of life assessment, and profile of mood states. Blood will be drawn at each study visit.

ELIGIBILITY:
Inclusion criteria

* HIV infection
* History of a CD4 cell count less than 200 cells/mm3
* Stable antiretroviral regimen
* English-speaking

Exclusion criteria

* Inability or unwillingness to fill out questionnaires
* History of non-HIV related life-threatening disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-12; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Donald Abrams, MD, Principal Investigator — University of California, San Francisco; Jerome J. Stone, MA, RN, Study Director — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States